CLINICAL TRIAL: NCT05890755
Title: Mimicking Slipping Responses Using a Novel Mechanical Perturbation Algorithm
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00213
Record Dates: First submitted 2023-03-31; First posted 2023-06-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Gait, Stumbling; Gait, Perturbation
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy participants between 18 and 40 years of age
  Interventions: Other: Mechanical pertubation
- Healthy participants between 60 and 80 years of age
  Interventions: Other: Mechanical pertubation

INTERVENTIONS:
Other: Mechanical pertubation — Acceleration or deacceleration of one treadmill gait belt.

SUMMARY:
Healthy subjects will be invited to fill out a questionnaire regarding falls and balance skills followed by normal walking trials on a treadmill at 9 different speeds (0.28-1.4 m/s). Key gait parameters for the normative database will be collected. During the perturbation trials, the subjects will walk at a constant speed (1.2 m/s). The treadmill belts are ac, - or decelerated during the perturbations according to three different perturbation algorithms with varying perturbation onset. Movements will be analyzed by 3D motion capture, force plates, surface electromyography and IMU sensors. All methods are non-invasive and commonly used in the field of biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18-40 years and 60-80 years
* Ability to walk at minimum 30 minutes at a regular pace without assistance or breaks
* Written informed consent as documented by signature (see informed consent form)

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Current neurological problems affecting walking function and balance
* Current orthopedic problems affecting upper and lower extremity movements
* History of alcohol abuse or the intake of psychotropic drugs
* History of major cardiac condition (e.g., infarction, insufficiency (NYHA II-IV))
* History of major pulmonary condition (e.g., chronic obstructive pulmonary disease (GOLD II-IV))
* Current major depression or psychosis
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia
* Fever of unknown origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy population
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Calculation of Margins of Stability (MoS) in anterior-posterior direction at foot contact | Once during visit 1
  Difference between base of support and interpolated center of mass (mm), based on 3D motion capture.
Step length at baseline, before (Pre) and after (Recovery step 1-10) perturbation | Once during visit 1

SECONDARY OUTCOMES:
Step width at foot contact of baseline, before (Pre) and Recovery steps 1-10 | Once during visit 1
Calculation of Margin of stability medial-lateral direction at foot contact of baseline, before (Pre) and Recovery steps 1-10 | Once during visit 1
  Difference between base of support and interpolated center of mass (mm), based on 3D motion capture.
Maximal trunk velocity during gait cycle at of baseline, before (Pre) and Recovery steps 1-10 to detect fast trunk movement to gain balance | Once during visit 1
  Optical markers are placed on the upper body of the subjects and will be used for calculation (distance over time) of the trunk velocity.
3D kinematic gait profiles to analyze detailed movement patterns/strategies | Once during visit 1
  The optical markers are placed according to the Plug-in gait marker set in Vicon Nexus (motion capture system). Hip, knee, ankle and trunk angles are calculated from this marker set.
EMG analysis to detect reaction time and activity patterns of different leg muscles | Once during visit 1
Questionnaire regarding the incidence of falls in the last six months | Once during visit 1
  Contains questions how often und the reason why the subject falls
Activities specific Balance Confidence scale (ABC scale) | Once during visit 1
  Contains 16 questions rating the balance confidence between 0-100%. 100% means absolutely confident in doing some activity
Questionnaire regarding the perceived intensities of the three perturbation algorithms | Once during visit 1
  Judging the three pertubation algorithms according to their intensity, inconvenience and how realistic the slipping felt. Scale ranges from 0-10, whereas 10 is the most intense
Functional Gait Assessment (FGA) as a clinical balance test | Once during visit 1
  Assess the dynamic stability during different walking tasks. In total, 30 points are possible, at 22 points is the cut off score to classify the fall risk in older adults in predicting falls.
A set of kinematic parameters | Once during visit 1
  Measurement of hip, knee, ankle and spine angles during walking in degrees (°).
A set of kinetic parameters | Once during visit 1
  Ground reaction forces measured by force plates in Newton (N).
A set of spatiotemporal parameters | Once during visit 1
  Stance time, double stance time in seconds (s).

CONTACTS AND LOCATIONS:
Overall Officials: Linard Filli, Dr., Principal Investigator — University of Zurich
Locations (1):
- Balgrist Campus, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No